CLINICAL TRIAL: NCT04604535
Title: The Effects of Dietary Nitrate Supplementation on Pregnancies Complicated by Chronic and New Onset Hypertension
Brief Title: The BEET-BP Trial - Investigating the Effect of Dietary Nitrates on Hypertension in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Fetal Medicine Foundation (Other); Barts and the London School of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263871
Record Dates: First submitted 2020-10-12; First posted 2020-10-27 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Hypertension in Pregnancy; Pre-Eclampsia; Gestational Hypertension; Pregnancy Induced Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated beetroot juice (Active Comparator): 70mL of concentrated beetroot juice with 400mg nitrate
  Interventions: Dietary Supplement: Concentrated beetroot juice
- Placebo (Placebo Comparator): 70mL of concentrated beetroot juice with <0.01mmol/L nitrate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Concentrated beetroot juice — 70mL concentrated beetroot juice (400mg nitrate)
  Arms: Concentrated beetroot juice
Dietary Supplement: Placebo — 70mL concentrated nitrate deplete beetroot juice (<0.01mmol/L nitrate)
  Arms: Placebo

SUMMARY:
This is a randomised placebo controlled trial investigating the effects of dietary nitrate supplementation on hypertension in pregnancy

DETAILED DESCRIPTION:
Reduced nitrate and nitrite concentrations have been found in women with preeclampsia (PE) and studies have shown increased concentrations of an endogenously generated Nitric Oxide Synthase inhibitor, amongst women with PE.

Nitrate and nitrite are required to produce Nitric Oxide (NO). NO is released from the endothelial lining of blood vessels, and acts to relax smooth muscle within the vasculature, acting as a potent vasodilator. Reduced NO concentrations are hence thought to contribute towards the systemic vascular constriction seen in PE.

Hypertensive diseases in pregnancy are an important cause of morbidity and mortality in both maternal, fetal and neonatal health. Treatment options are limited in pregnancy and hence alternative methods to improve blood pressure control should be sought.

In this randomised placebo controlled double blinded trial we aim to assess the effect of dietary nitrate supplementation on the hypertensive diseases of pregnancy and the subsequent maternal, fetal-neonatal outcomes. The safety and acceptability of dietary nitrate supplementation will also be confirmed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Able to give written informed consent
* Singleton pregnancies, between 24+0 to 36+6 weeks gestation with new onset gestational hypertension (defined by ISSHP2018 as new onset BP >140/90 and no evidence of proteinuria, biochemical or haematological abnormalities or fetal growth restriction) Or
* Singleton pregnancies, between 24+0 - 36+6 weeks gestation, with chronic hypertension (defined by ISSHP2018 as BP ≥140/90 predating the pregnancy or recognised at <20 week's gestation) Or
* Singleton pregnancies, between 24+0 - 36+6 weeks gestation, with preeclampsia (defined by ISSHP2018 as Gestational hypertension accompanied by ≥ 1 of the following new onset conditions at or after 20 weeks' gestation:
* Proteinuria (24h urine collection>300mg/day, Protein-creatinine ratio>30 mg/mmol)
* Other markers of maternal organ dysfunction, including:
* Acute Kidney Injury (AKI) (creatinine ≥90μmol/L; 1mg/dL)
* Liver involvement (elevated transaminases e.g. alanine transaminase (ALT) or aspartate aminotransferase (AST) >40IU/L) with or without right upper quadrant or epigastric abdominal pain
* Neurological complications e.g. eclampsia, altered mental status, blindness, stroke, clonus, severe headaches and persistent visual scotomata
* Haematological complications (thrombocytopenia - platelet count <150 000/μL, disseminated intravascular coagulation, haemolysis
* Uteroplacental dysfunction (fetal growth restriction, abnormal umbilical artery doppler wave form analysis, or stillbirth)

Exclusion Criteria:

* Unable to tolerate taste of beetroot juice concentrate during taste test
* Multiple pregnancy
* History of acute or chronic liver conditions (aside from preeclampsia)
* Fetal aneuploidies or major fetal anomalies
* Unwillingness to comply with all study-related procedures e.g. Women who have used mouthwash or tongue scraping in last 7 days and are not able/unwilling unable to stop this for the duration of the study
* Women on treatment for gingivitis
* Women with persistent hyperemesis or ptyalism
* On Proton-pump-inhibitors/antacids other treatment for gastritis/peptic ulcer/gastric ulcers
* Those with long term antibiotic use e.g. prophylaxis of urinary tract infections (UTIs) or those who are likely to need repeated courses of antibiotics e.g. history of recurrent UTI
* Women with known allergy/intolerance to beetroot or lemon
* Type 1 and Type 2 diabetics
* Moderate iron deficiency anaemia with haemoglobin <100g/dL and/or ferritin <15μg/L
* Any blood disorder or significant illness that may affect platelet function and coagulation. However, patients taking low-dose aspirin (150mg) for preeclampsia prophylaxis who are at increased risk of developing preeclampsia will be included in the study.
* History of alcohol or recreational drug abuse use within the past 6 months
* Systemic autoimmune disease e.g. Rheumatoid Arthritis, antiphospholipid syndrome connective tissue disease e.g. Systemic Lupus Erythematous or other conditions known to be associated with chronic inflammation such as inflammatory bowel disease - Chron's disease/Ulcerative Colitis
* Women not intending to deliver at the recruiting site
* Participating in another intervention study that influences the outcomes of this study
* Those with serious mental illness or learning difficulties and unable to give written informed consent
* Those who are detained as a prisoner or detained in any secured unit, including those held under the Mental Health Act
* Those not fluent in local language, and absence of appropriate interpreter despite use of services such as Language Line

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-10-22 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Gestational age of delivery secondary to preeclampsia | From recruitment until delivery

SECONDARY OUTCOMES:
Gestational age of delivery (due to any cause) | From recruitment until delivery
Will beetroot juice supplementation increase or decrease the likelihood of maternal complications, including severe maternal complications | From recruitment until 8 weeks postnatal
Will beetroot juice supplementation increase or decrease the likelihood of severe hypertension | From recruitment until 8 weeks postnatal
  Defined as ≥ 160/110 mmHg
Will beetroot juice supplementation result in significant changes in systolic blood pressure and diastolic blood pressure | From recruitment until 8 weeks postnatal
Will beetroot juice supplementation result in a significant change in the maximal number and dosages of antihypertensive medications required for blood pressure control | From recruitment until 8 weeks postnatal
Will beetroot juice supplementation result in a significant change in maternal blood values and urinary protein excretion | From recruitment until 8 weeks postnatal
  Measured by creatinine, aspartate aminotransferase, alanine aminotransferase, uric acid, platelets, random urine protein creatinine ratio, protein concentration in a 24hour urine collection
Can the safety of beetroot juice supplementation in pregnancy be confirmed | From recruitment until 8 weeks postnatal
  Measurement of maternal methemoglobinaemia levels, maternal nitrosamine levels, maternal thyroid function, neonatal cord bloods, neonatal methemoglobinaemia levels
To confirm the acceptability of beetroot juice supplementation in pregnancy | At 8 weeks postnatal
  A post-trial questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nick Kametas, Study Chair — Fetal Medicine Research Institute, King's College Hospital London; Kypros Nicolaides, Study Chair — Fetal Medicine Research Institute, King's College Hospital London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No